CLINICAL TRIAL: NCT01604278
Title: A 12-week Multi-center, Randomized, Double-blind, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of the Co-administration of NVA237 + Indacaterol Once Daily vs. Indacaterol Once Daily in Patients With Moderate to Severe COPD
Brief Title: Efficacy, Safety and Tolerability of the Co-administration of NVA237 Plus Indacaterol Once Daily Versus Indacaterol Once Daily in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Acronym: GLOW6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNVA237A2316; 2011-005673-23 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Indacaterol; Glycopyrronium Bromide; COPD; bronchodilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- NVA237 + indacaterol (Active Comparator)
  Interventions: Drug: NVA237 50 µg and indacaterol 150 µg
- Placebo to NVA237 + indacaterol (Placebo Comparator)
  Interventions: Drug: Placebo to NVA237 and indacaterol 150 µg

INTERVENTIONS:
Drug: NVA237 50 µg and indacaterol 150 µg — NVA237 50 µg and indacaterol 150 µg supplied as blistered capsules for inhalation.
  Other Names: Glycopyrronium Bromide
  Arms: NVA237 + indacaterol
Drug: Placebo to NVA237 and indacaterol 150 µg — Placebo to NVA237 and indacaterol 150 µg supplied as blistered capsules for inhalation.
  Arms: Placebo to NVA237 + indacaterol

SUMMARY:
This study assessed the efficacy, safety and tolerability of the co-administration of NVA237 plus indacaterol taken once daily versus indacaterol taken once daily in patients with moderate to severe Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe stable Chronic Obstructive Lung Disease (COPD) Stage II or Stage III according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines.
* Patients with a post-bronchodilator forced expiratory volume in 1 second (FEV1) ≥ 30 % and/or <80 % of the predicted normal, and a post-bronchodilator FEV1/Forced Vital Capacity (FVC) < 0.70 at screening.
* Current or ex-smokers who have a smoking history of at least 10 pack years
* Symptomatic patients according to daily diary data.

Exclusion Criteria:

* Pregnant or nursing (lactating) women.
* Women of child-bearing potential unless using adequate contraception.
* Patients with Type I or uncontrolled Type II diabetes.
* Patients with a history of long time interval between start of Q wave and end of T wave in the heart's electrical cycle (QT) syndrome or whose QT corrected for heart rate (QTc) measured at screening (Visit 2) (Fridericia's method) is prolonged
* Patients with paroxysmal (e.g. intermittent) atrial fibrillation
* Patients who have a clinically significant electrocardiogram (ECG) or laboratory abnormality at screening (Visit 2)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- Belgium (13):
  - Novartis Investigative Site, Malmedy/Bellevaux-Ligneuville, Belgium
  - Novartis Investigative Site, Luxembourg, Luxembourg
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Gilly
  - Novartis Investigative Site, Gosselies
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Herentals
  - Novartis Investigative Site, Jambes
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Montigny-le-Tilleul
  - Novartis Investigative Site, Turnhout
  - Novartis Investigative Site, Yvoir
- Bulgaria (6):
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Stara Zagora
- Greece (3):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (4):
  - Novartis Investigative Site, Érd, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Gödöllő
- Novartis Investigative Site, Wilton, Cork, Ireland
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Saratov
- Slovakia (7):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Kráľovský Chlmec, Slovakia
  - Novartis Investigative Site, Námestovo, Slovensko
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- Spain (11):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Torrelavega, Cantabria
  - Novartis Investigative Site, Ponferrada, Castille and León
  - Novartis Investigative Site, Illescas, Castille-La Mancha
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Salt, Catalonia
  - Novartis Investigative Site, Sant Boi de Llobregat, Catalonia
  - Novartis Investigative Site, Viladecans, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Gijón, Principality of Asturias
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Yenisehir/Izmir
- United Kingdom (20):
  - Novartis Investigative Site, Burnhope, County Durham
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle-upon-Tyne
  - Novartis Investigative Site, Alderton, Suffolk
  - Novartis Investigative Site, Cambridge, United KIngdom
  - Novartis Investigative Site, Watford, United Kingdom
  - Novartis Investigative Site, Atherstone, Warwickshire
  - Novartis Investigative Site, Royal Leamington Spa, Warwickshire
  - Novartis Investigative Site, Strensall, Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Bexhill-on-Sea
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Huntingdon
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newton Aycliffe
  - Novartis Investigative Site, Reading
  - Novartis Investigative Site, Southbourne
  - Novartis Investigative Site, Telford
  - Novartis Investigative Site, Wiltshire

REFERENCES:
- [Derived] Vincken W, Aumann J, Chen H, Henley M, McBryan D, Goyal P. Efficacy and safety of coadministration of once-daily indacaterol and glycopyrronium versus indacaterol alone in COPD patients: the GLOW6 study. Int J Chron Obstruct Pulmon Dis. 2014 Feb 24;9:215-28. doi: 10.2147/COPD.S51592. eCollection 2014. PMID 24596459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of patients randomized was 449. Of these participants, the Full Analysis Set (FAS) comprised 446 participants who received at least one dose of study drug and had no major deviations which led to removal from the FAS. The Safety Set included 447 participants who received at least one dose of study drug.
Groups:
- NVA237 + Indacaterol: Participants received Indacaterol 150 ug once daily delivered via single dose dry powder inhaler (SDDPI) plus NVA237 50 ug once daily delivered via SDDPI
- Placebo to NVA237 + Indacaterol: Participants received Indacaterol 150 ug once daily delivered via SDDPI plus placebo to NVA237 delivered via SDDPI
Period: Overall Study
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Started | 226 | 223
Safety Set | 226 | 221 (Two randomized participants who did not receive study drug were excluded from this set.)
Full Analysis Set | 226 | 220 (Three randomized participants excluded: 2 who did not receive study drug; 1 with a major deviation.)
Completed | 212 | 210
Not Completed | 14 | 13
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Adverse Event | 3 | 5
Not completed — Protocol Deviation | 5 | 3

BASELINE CHARACTERISTICS:
Population: The baseline characteristics table was based on the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol | Total
Number analyzed (Participants) | 226 | 221 | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.44) | 64.1 (7.67) | 63.7 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 35 | 81
  Male | 180 | 186 | 366

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume at 1 Second (FEV1)
Description: Centralized spirometry according to internationally accepted standards was used. The model contained treatment, baseline smoking status and baseline inhaled corticosteroid (ICS) use as fixed effects with the baseline measurement of FEV1, FEV1 prior to inhalation of short acting bronchodilators and FEV1 post inhalation of short acting bronchodilator as covariates and center nested in region as a random effect. If trough FEV1 was missing at week 12, the latest non-missing pre-dose trough FEV1 (the mean of 45 and 15 min pre-dose measurements) from day 29, 57 or 84) was carried forward. These measurements had to have been taken before the next dose of study medication. FEV1 measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were not included in the analysis.
Time Frame: 12 weeks
Population: Only participants from the full analysis set, who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 214 | 214
Liters | 1.499 (0.0135) | 1.436 (0.0136)

2. Secondary Outcome: FEV(1) Area Under the Curve (AUC) During 30 Minutes to 4 Hours Post Dose
Description: Centralized spirometry was used according to internationally accepted standards was used. The trapezoidal rule was applied to calculate FEV1 Area Under the Curve (AUC) and then normalized to the length of time. Whether the participants had complete or incomplete FEV1 assessments in respective time ranges, their AUCs were calculated based on the existing FEV1 measurements (i.e., the missing FEV1 measurements were not interpolated). Specifically, for those participants who had a FEV1 assessment at only one time-point, their AUC was approximated by the observed FEV1. FEV1 measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were not included in the analysis.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 208 | 208
Liters | 1.641 (0.0132) | 1.530 (0.0134)

3. Secondary Outcome: Peak FEV1 During 30 Minutes to 4 Hours Post-dose at 12 Weeks
Description: Centralized spirometry was used according to internationally accepted standards was used. Peak FEV1 was defined as the maximum FEV1 during the first 4 hours post morning dosing. The model contained treatment, baseline smoking status and baseline ICS use as fixed effects with the baseline measurement of FEV1, FEV1 prior to inhalation of short acting bronchodilators and FEV1 post inhalation of short acting bronchodilator as covariates and center nested in a region as a random effect. If all FEV1 measurements were missing from 30 minutes onward, the peak FEV1 was not calculated. FEV1 measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were not included in the analysis.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 208 | 208
Liters | 1.702 (0.0137) | 1.596 (0.0138)

4. Secondary Outcome: FEV1 at Individual Time-points
Description: Centralized spirometry according to internationally accepted standards was used. FEV1 was measured at all post-dose time points up to 4 hours, and at 23 hours 15 minutes and 23 hours 45 minutes, by visit. The model contained treatment, baseline smoking status and baseline ICS use as fixed effects with the baseline measurement of FEV1, FEV1 prior to inhaltion of short acting bronchodilators and FEV1 post inhaltion of short acting bronchodilators as covariates and center nested in region as a random effect. FEV1 measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were not included in the analysis.
Time Frame: Day 1, Day 29, Day 57 and Days 84/85
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 226 | 220
Liters
  Day 1, 30 minutes (min) post dose (n=208,199) | 1.544 (0.0086) | 1.467 (0.0088)
  Day 1, 1 hour (h) post dose (n=214,209) | 1.589 (0.0102) | 1.479 (0.0104)
  Day 1, 2 h post dose (n=212,207) | 1.626 (0.0114) | 1.506 (0.0117)
  Day 1, 4 h post dose (n=206,213) | 1.630 (0.0122) | 1.518 (0.0122)
  Day 1, 23 h 15 min post dose (n=201,203) | 1.481 (0.0118) | 1.409 (0.0118)
  Day 1, 23 h 45 min post dose (n=213,204) | 1.502 (0.0109) | 1.425 (0.0112)
  Day 29, 45 min pre-dose (n=198,202) | 1.491 (0.0150) | 1.438 (0.0150)
  Day 29, 15 min pre-dose (n=198,200) | 1.524 (0.0156) | 1.470 (0.0155)
  Day 29, 30 min post dose (n=202,201) | 1.617 (0.0152) | 1.508 (0.0154)
  Day 29, 1 h post dose (n=200,199) | 1.648 (0.0144) | 1.524 (0.0145)
  Day 56, 45 min pre-dose (n=201,202) | 1.482 (0.0145) | 1.418 (0.0146)
  Day 56, 15 min pre-dose (n=199,198) | 1.509 (0.0148) | 1.443 (0.0149)
  Day 56, 30 min post dose (n=200,200) | 1.606 (0.0144) | 1.495 (0.0146)
  Day 56, 1 h post dose (n=197,204) | 1.634 (0.0149) | 1.520 (0.0148)
  Days 84/85, 45 min pre-dose (n=201,206) | 1.459 (0.0127) | 1.411 (0.0126)
  Days 84/85, 15 min pre-dose (n=190,196) | 1.476 (0.0129) | 1.439 (0.0129)
  Days 84/85, 30 min post dose (n=198,199) | 1.604 (0.0125) | 1.514 (0.0126)
  Days 84/85, 1 h post dose (n=201,200) | 1.638 (0.0125) | 1.514 (0.0126)
  Days 84/85, 2 h post dose (n=198,201) | 1.665 (0.0139) | 1.542 (0.0139)
  Days 84/85, 4 h post dose (n=200,198) | 1.620 (0.0162) | 1.529 (0.0165)
  Days 84/85, 23 h 15 min post dose (n=193,188) | 1.474 (0.0139) | 1.426 (0.0143)
  Days 84/85, 23 h 45 min post dose (n=197,199) | 1.508 (0.0147) | 1.452 (0.0148)

5. Secondary Outcome: Forced Vital Capacity (FVC) at Individual Time-points
Description: FVC was calculated at each time point up to 4 hours post-dose and at 23 hours 15 minutes and 23 hours 45 minutes, by visit. The model contained treatment, baseline smoking status and baseline ICS use as fixed effects with the baseline measurement of FVC, FEV1 prior to inhaltion of short acting bronchodilators and FEV1 post inhaltion of short acting bronchodilators as covariates and center nested in region as a random effect. FVC measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were set to missing.
Time Frame: Day 1, Day 29, Day 57 and Days 84/85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 226 | 220
Liters
  Day 1, 30 min post dose (n=208,199) | 3.214 (0.0181) | 3.135 (0.0186)
  Day 1, 1 h post dose (n=214,209) | 3.295 (0.0260) | 3.182 (0.0264)
  Day 1, 2 h post dose (n=212,207) | 3.325 (0.0229) | 3.200 (0.0234)
  Day 1, 4 h post dose (n=206,213) | 3.340 (0.0239) | 3.218 (0.0238)
  Day 1, 23 h 15 min post dose (n=201,203) | 3.155 (0.0267) | 3.039 (0.0268)
  Day 1, 23 h 45 min post dose (n=213,204) | 3.201 (0.0257) | 3.095 (0.0263)
  Day 29, 45 min pre-dose (n=198,202) | 3.146 (0.0299) | 3.043 (0.0299)
  Day 29, 15 min pre-dose (n=198,200) | 3.184 (0.0315) | 3.092 (0.0314)
  Day 29, 30 min post dose (n=202,201) | 3.316 (0.0338) | 3.201 (0.0341)
  Day 29, 1 h post dose (n=200,199) | 3.362 (0.0336) | 3.197 (0.0337)
  Day 56, 45 min pre-dose (n=201,202) | 3.102 (0.0302) | 3.015 (0.0303)
  Day 56, 15 min pre-dose (n=199,198) | 3.156 (0.0321) | 3.086 (0.0322)
  Day 56, 30 min post dose (n=200,200) | 3.282 (0.0316) | 3.190 (0.0319)
  Day 56, 1 h post dose (n=197,204) | 3.327 (0.0323) | 3.219 (0.0321)
  Days 84/85, 45 min pre-dose (n=201,206) | 3.052 (0.0280) | 3.016 (0.0279)
  Days 84/85, 15 min pre-dose (n=190,196) | 3.064 (0.0256) | 3.012 (0.0254)
  Days 84/85, 30 min post dose (n=198,199) | 3.246 (0.0262) | 3.162 (0.0264)
  Days 84/85, 1 h post dose (n=201,200) | 3.312 (0.0291) | 3.179 (0.0294)
  Days 84/85, 2 h post dose (n=198,201) | 3.318 (0.0261) | 3.181 (0.0261)
  Days 84/85, 4 h post dose (n=200,198) | 3.251 (0.0292) | 3.161 (0.0297)
  Days 84/85, 23 h 15 min post dose (n=193,188) | 3.123 (0.0285) | 3.050 (0.0292)
  Days 84/85, 23 h 45 min post dose (n=197,199) | 3.136 (0.0256) | 3.047 (0.0258)

6. Secondary Outcome: Inspiratory Capacity (IC) at Individual Time-points
Description: Inspiratory Capacity (IC) was measured at 20 min pre-dose and at post-dose at 25 minutes, 1 hour 55 minutes, 3 hours 55 minutes and 23 hours 40 minutes, by visit. The model contained treatment, baseline smoking status and baseline ICS use as fixed effects with the baseline measurement of IC, FEV1 prior to inhalation of short acting bronchodilators and FEV1 post inhalation of short acting bronchodilators as covariates and center nested in region as a random effect. IC measurements within 6 hours of rescue medication use or within 7 days of systemic corticosteroid use were set to missing.
Time Frame: Day 1, Days 84/85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 226 | 220
Liters
  Day 1, 25 min post dose (n=164,168) | 2.493 (0.0234) | 2.434 (0.0231)
  Day 1, 1 h 55 min (n=161,176) | 2.587 (0.0294) | 2.478 (0.0287)
  Day 1, 3 h 55 min (n=160,173) | 2.557 (0.0298) | 2.475 (0.0291)
  Days 84/85, 20 min pre-dose (n=144,148) | 2.444 (0.0327) | 2.363 (0.0324)
  Days 84/85, 25 min post dose (n=149,145) | 2.580 (0.0372) | 2.420 (0.0377)
  Days 84/85, 1 h 55 min post dose (n=146,153) | 2.607 (0.0388) | 2.485 (0.0384)
  Days 84/85, 3 h 55 min (n=146,145) | 2.577 (0.0332) | 2.439 (0.0333)
  Days 84/85, 23 h 40 min (n=153,150) | 2.405 (0.0371) | 2.337 (0.0376)

7. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication
Description: The number of puffs of rescue medication taken in the previous 12 hours was recorded in the patient diary in the morning and evening. The total number of puffs of rescue medication per day over the whole active treatment period was calculated and divided by the total number of days with non-missing rescue data to derive the mean daily number of puffs of rescue medication taken for the patient. If the number of puffs was missing for part of the day (either morning or evening), then a half day was used in the denominator.
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 219 | 216
Number of puffs | -1.9 (0.16) | -1.8 (0.16)

8. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score
Description: Dyspnea was measured at baseline using the Baseline Dyspnea Index (BDI) and during treatment using the Transitional Dyspnea Index (TDI). Analysis was done via mixed model. The BDI and TDI each have three domains: functional impairment, magnitude of task and magnitude of effort. BDI domains were rated from 0 (severe) to 4 (unimpaired) and rates summed for baseline focal score ranged from 0 to 12; lower scores mean worse severity. TDI domains were rated from -3 (major deterioration) to 3 (major improvement) and rates summed for transition focal score ranged from -9 to 9; negative scores indicate deterioration. A TDI focal score of 1 is considered a minimal clinically important difference.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 207 | 209
Score | 2.506 (0.2781) | 2.012 (0.2797)

9. Secondary Outcome: Change From Baseline in Mean Daily Total and Individual Symptom Scores
Description: The symptoms (respiratory, cough, wheeze, sputum color, sputum production, breathlessness, sore throat, nasal discharge or congestion, and fever) for the whole active treatment period was analyzed using a mixed model, which contained treatment, baseline smoking status and baseline ICS use as fixed effects with the baseline symptom score, FEV1 prior to inhalation of short acting bronchodilators and FEV1 post inhalation of short acting bronchodilators as covariates and center nested in region as a random effect. Each symptom was scored as 0, 1, 2 or 3 where the description for each score varied. For each of the symptoms, the range of scores from 0 to 3 represented an increase in symptoms where 0 represented little to no symptom and 3 represented severe or worst symptom. The total symptom score, which is the sum of the individual scores, ranged from 0 (best possible outcome) to 27 (worst possible outcome).
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 212 | 214
Score
  Total symptom score | -1.2 (0.13) | -1.1 (0.13)
  Respiratory symptom score | -0.3 (0.03) | -0.2 (0.03)
  Cough symptom score | -0.2 (0.03) | -0.2 (0.03)
  Wheeze symptom score | -0.3 (0.03) | -0.2 (0.03)
  Sputum production score | -0.1 (0.03) | -0.1 (0.03)
  Sputum color score | -0.1 (0.02) | -0.1 (0.02)
  Breathless symptom score | -0.2 (0.03) | -0.2 (0.03)
  Sore throat symptom score | 0.0 (0.01) | 0.0 (0.01)
  Cold symptom score | 0.0 (0.02) | 0.0 (0.02)
  Fever symptom score | 0.0 (0.01) | 0.0 (0.01)

10. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: All study emergent adverse events including Chronic Obstructive Pulmonary Disease exacerbations were monitored from screening through the end of study.
Time Frame: 12 weeks
Population: Safety Set: The safety set included all patients who received at least one dose of study drug whether or not they were randomized.
Measure: Number; unit: Number of participants
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Number analyzed (Participants) | 226 | 221
Number of participants
  Adverse Events (serious and non-serious) | 85 | 75
  Serious adverse events | 5 | 5
  Deaths | 0 | 0

ADVERSE EVENTS:
Arm/Group | NVA237 + Indacaterol | Placebo to NVA237 + Indacaterol
Serious Adverse Events (participants affected / at risk) | 5/226 | 5/221
Other Adverse Events (participants affected / at risk) | 32/226 | 27/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 + Indacaterol (N=226) | Placebo to NVA237 + Indacaterol (N=221)
Angina pectoris (Cardiac disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 + Indacaterol (N=226) | Placebo to NVA237 + Indacaterol (N=221)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 32 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.